CLINICAL TRIAL: NCT05719935
Title: The KinematX Midcarpal Total Wrist Arthroplasty: A Multicenter Prospective Registry of Clinical and Patient-Reported Outcomes
Brief Title: The KinematX Midcarpal Total Wrist Arthroplasty Registry
Status: Recruiting | Type: Observational
Sponsor: Extremity Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 112020-1
Record Dates: First submitted 2022-12-19; First posted 2023-02-09 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Scapholunate Advanced Collapse (SLAC); Scapholunate Crystalline Advanced Collapse (SCAC); Scaphoid, Trapezium, and Trapezoid Advanced Collapse (STTAC); Carpal Tunnel Syndrome (CTS); Kienbock's Disease of Adults; Radial Malunion; Ulnar Translocation; Post Traumatic Arthritis; Inflammatory Arthritis; Osteoarthritis; Scaphoid Non-union Advanced Collapse (SNAC)
Keywords: Total wrist replacement; Total wrist arthroplasty
MeSH Terms: conditions — Carpal Tunnel Syndrome; Arthritis; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- KinematX patients: Patients undergoing total wrist replacement with the KinematX implant.
  Interventions: Device: KinematX total wrist arthroplasty system

INTERVENTIONS:
Device: KinematX total wrist arthroplasty system — The KinematX total wrist implant is a joint metal/polymer semi-constrained cemented prosthesis that utilizes an articulation that mimics the midcarpal joint instead of the radiocarpal joint.

SUMMARY:
The goal of this observational study is to learn about functional and patient reported outcomes in patient undergoing total wrist replacement with the KinematX total wrist replacement study.

The main questions it aims to answer are:

* What is the range of motion (flexion, extension, radial, ulnar, grip and pinch strength) at 3-, 6-, and 12-months after surgery and yearly up to 10 years among patients having total wrist replacement with the KinematX implant.
* What are the patient reported outcomes (PROMIS, PRWE, HSS wrist expectations) at 3-, 6-, and 12-months after surgery and yearly up to 10 years among patients having total wrist replacement with the KinematX implant.
* How do range of motion and patient reported outcomes change over the 10 years after total wrist replacement surgery?

Participants will be followed according to standard of care and preoperative and post-operative information for up to 10 years after surgery will be collected and entered into an electronic data base. Patients are eligible to enroll into the registry before or after they have had their wrist replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* one of the following diagnoses and planned (or previously completed) total wrist arthroplasty with the KinematX total wrist:

  * osteoarthritis or post-traumatic arthritis
  * scapholunate advanced collapse (SLAC/SNAC wrist),
  * inflammatory arthritis (rheumatoid, psoriatic, other),
  * crystalline advanced collapse (SCAC),
  * STT advanced collapse (STTAC),
  * ulnar translocation,
  * Kienbӧck disease,
  * radial malunion

Exclusion Criteria:

* <18 years of age
* >85 years of age
* Prisoners
* Children
* Pregnant women
* Contraindications to receiving the KinematX:

  * Local, distant or systematic acute or chronic soft tissue or bony infection
  * Physiologically or psychologically compromised patient
  * Active wrist synovitis or severe carpal bone erosion
  * Suspected or documented metal allergy or intolerance
  * Insufficient extensor tendons
  * Inadequate skin, bone, neural or vascular status
  * Severe carpal bone malalignment, displacement, absorption, neoplastic, or carpal bone pathology
  * Sepsis
  * Osteomyelitis
  * Uncontrolled/untreated osteoporosis or metabolic bone disease
  * Metabolic or endocrinologic bone disorders
  * Osteomalacia
  * Distant foci of infections which may spread to the implant site
  * Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-85 with planned (or previously completed) total wrist arthroplasty with the KinematX total wrist are eligible for enrollment into this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Range of Motion (as assessed by physician) | Up to 10 years
  Flexion, Extension, Ulnar, Radial

SECONDARY OUTCOMES:
PROMIS Upper Extremity Physical Function 7a | 3 months, 6 months, yearly up to 10 years post-surgery
  7 questions designed to understand the patient's physical function in the upper extremity specifically; population average t-score is 50, with a standard deviation of 10; higher scores are better.
PROMIS Pain Interference 8a | 3 months, 6 months, yearly up to 10 years post-surgery
  8 questions designed to understand how any pain experienced interferes with the patient's day to day life; population average t-score is 50, with a standard deviation of 10; lower scores are better
PROMIS Global 10 | 3 months, 6 months, yearly up to 10 years post-surgery
  10 questions to assess the patient's global health with subscales for physical health and mental health; Physical health t-scores range from 16.2 to 67.7; Mental health t-scores range from 21.2 to 67.6; higher scores are better
Patient-Rated Wrist Evaluation Score (PRWE) | 3 months, 6 months, yearly up to 10 years post-surgery
  15 questions that assess pain and function; total scores can range from 0-100; lower scores are better
Hospital for Special Surgery Wrist Surgery Expectations Survey | Pre-operative and yearly up to 10 years post-surgery
  22 questions that assess how the patient expects to benefit from the surgery and a corresponding post-operative instrument that asks about actual experience; score range from 22 to 110; lower scores are better
Percentage of patients experiencing post-operative complications | 3 months, 6 months, yearly up to 10 years post-surgery
Percentage of patients requiring revision surgery for their implant (with or without implant replacement) | 3 months, 6 months, yearly up to 10 years post-surgery
Grip and pinch strength (as assessed by physician) | 3months, 6 months, yearly up to 10 years post-surgery
  Grip and pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Brian Smekal, Study Director — Extremity Medical
Locations (4):
- United States (4):
  - Loma Linda University, Loma Linda, California
  - Florida Orthopaedic Institute, Tampa, Florida
  - Franciscan Health, Indianapolis, Indiana
  - Hospital for Special Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No